CLINICAL TRIAL: NCT04826783
Title: Effect of Various Laser Systems in Smokers and Nonsmokers With Peri-implantitis: A Randomized, Prospective, Single-Blind Clinical Trial
Brief Title: Use of Various Laser Systems in Peri-implatit
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kırıkkale University (Other)
Responsible Party: Principal Investigator, Kubilay BARIŞ, dr., Kırıkkale University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Interventional
Record Dates: First submitted 2021-01-23; First posted 2021-04-01 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: Peri-Implantitis
MeSH Terms: conditions — Peri-Implantitis | interventions — Lasers

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Diode laser (Experimental)
  Interventions: Device: Lasers
- Er,Cr:YSGG laser (Experimental)
  Interventions: Device: Lasers
- Er:YAG LAser (Experimental)
  Interventions: Device: Lasers

INTERVENTIONS:
Device: Lasers — The laser tip was applied as vertical and horizontal scan along the subgingival implant . The procedure was carried out on day zero, seven and 14.

SUMMARY:
Objectives: In recent years, a new field of work has been created with the use of laser beam to provide titanium surface decontamination. The aim of this study was to evaluate the effect of various laser systems in smokers and non-smokers with peri-implantitis.

Materials and Methods: According to the study protocol, patients, who were diagnosed with peri-implantitis based on the clinical and radiographic evaluations, were divided into six groups: Group 1: smokers undergoing diode laser application; Group 2: smokers undergoing Erbium, chromium: yttrium, scandium, gallium, garnet (Er, Cr:YSGG) laser application; Group 3: smokers undergoing Erbium:yttrium-aluminum-garnet (Er:YAG) laser application; Group 4: non-smokers undergoing diode laser application; Group 5: non-smokers undergoing Er, Cr:YSGG laser application; and Group 6: non-smokers undergoing Er:YAG laser application. Peri-implant sulcus depth (SD), clinical attachment level (CAL), suppuration, modified plaque index (mPI), gingival index (GI), and modified sulcus bleeding index (mSBI) were recorded and peri-implant sulcus fluid (PISF) was collected to evaluate osteocalcin.

ELIGIBILITY:
Inclusion Criteria:

1. Presence of pocket in probing depth of ≥4 mm in at least one implant
2. No mobility in implant
3. Implants with bridge foot and opposite occlusion
4. Having no systemic disease that may affect the outcome of treatment
5. No systemic use of antibiotics for the last six months
6. Not receiving peri-implantitis treatment for the last three months
7. Individuals at the 30-60 years of age.

Exclusion Criteria:

1. Individuals who did not agree to participate in the study
2. Individuals receiving radiation therapy
3. Individuals using alcohol
4. Presence of pregnancy and lactation period
5. Individuals with parafunctional habits such as clenching or bruxism.

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-04-25 (Estimated); Primary Completion 2021-10-25 (Estimated); Study Completion 2022-04-25 (Estimated)

PRIMARY OUTCOMES:
Sulcus depth | basaline - six month

CONTACTS AND LOCATIONS:
Locations (1):
- Kırıkkale University faculty of Dentistry, Yahşihan, Kırıkkale, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided